CLINICAL TRIAL: NCT04535102
Title: POLATUZUMAB PLUS BENDAMUSTINE PLUS RITUXIMAB (POLA+BR) AS SALVAGE THERAPY PRIOR TO AUTOLOGOUS STEM CELL TRANSPLANT FOR PATIENTS WITH RELAPSED OR PRIMARY REFRACTORY DIFFUSE LARGE B-CELL LYMPHOMA
Brief Title: POLA+BR for Relapsed or Refractory DLBCL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of sufficient patient population
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-1195.cc; P30CA046934 (NIH)
Record Dates: First submitted 2020-07-23; First posted 2020-09-01 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — polatuzumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Polatuzumab + BR (minimum 3 cycles) (Experimental): Patients will be treated with a minimum of 3 cycles up to a maximum six cycles to optimize response prior to ASCT (stem cell transplant) per investigator discretion
  Interventions: Drug: Polatuzumab Vedotin

INTERVENTIONS:
Drug: Polatuzumab Vedotin — Polatuzumab vedotin is an ADC designed for the targeted delivery of MMAE(mono-methyl auristatin E), a potent microtubule inhibitor to lymphoma cells expressing CD79b. MMAE has a mechanism of action that is similar to that of vincristine.

SUMMARY:
This is a phase II multicenter, open-label study of polatuzumab vedotin administered by IV infusion in combination with standard doses of bendamustine (B) and rituximab (R) in transplant-eligible patients with relapsed or refractory DLBCL. A total of 22 patients will be enrolled over a period of 2 years through the University of Colorado and additional study sites if applicable. Study treatment will be given in 21-day cycles for patients with DLBCL.

DETAILED DESCRIPTION:
The first day of treatment will constitute Cycle 1 Day 1. Patients will be treated with a minimum of three cycles and up to a maximum of 6 cycles to optimize responses prior to ASCT based on investigator discretion.

All patients will be evaluated for safety and efficacy according to the schedules of assessments.

All patients will be assessed for response to treatment by the investigator with the use of standard criteria according to the Modified Lugano Response Criteria at the following time points:

* At the time of screening
* At the time of primary response assessment (3 weeks after completion of study treatment (i.e., 3 weeks after Cycle 3 Day 1 or after last dose of study medication)

Imaging at these timepoints must include FDG-PET (18F-fluorodeoxyglucose-positron emission tomography) and a diagnostic-quality CT scan with both oral and IV contrast. A combined PET/CT scan is encouraged if feasible. CT scans with oral and IV contrast should include neck, chest, abdomen, and pelvic scans. In patients for whom contrast is contraindicated, (e.g., patients with contrast allergy or impaired renal clearance or patient denial), PET-CT scans without contrast are permitted so long as they permit consistent and precise measurement of target lesions during the study treatment period.

Patients will also be evaluated every 3 months for 2 years, or until disease progression, death, withdrawal of consent, or initiation of another anti-cancer therapy. Tumor assessments should also be performed to confirm clinical suspicion of relapse or disease progression for documentation. The study will end when all patients enrolled have been followed until death, have withdrawn consent, have been lost to follow-up, until 2-year follow up, or the Sponsor-investigator decides to end the trial, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Signed ICF
2. Age ≥ 18 years
3. Able to comply with the study protocol, in the investigator's judgment
4. Histologically confirmed DLBCL (Obtaining pathology samples is not required prior to enrollment, but confirmation of availability is required prior to enrollment)
5. Must have received at least one prior rituximab containing chemotherapy therapy for DLBCL.
6. Patients must be transplant-eligible and have either relapsed or have become refractory to a prior regimen.
7. The following DLBCL histologies would be considered eligible for study entry:

   o DLBCL, not otherwise specified (NOS) (including both GCB type and ABC type)
   * T-cell/histiocyte-rich large B-cell lymphoma
   * High-grade B-cell lymphoma with MYC and BCL-2 and/or BCL-6 rearrangements
   * High grade B-cell lymphoma, NOS
   * Primary mediastinal (thymic) large B-cell lymphoma
   * Epstein Barr virus positive DLBCL, NOS
   * HHV8-positive DLBCL, NOS
   * HIV positive DLBCL
8. At least one bi-dimensionally measurable lesion on imaging scan defined as > 1.5 cm in its longest dimension
9. Life expectancy of at least 24 weeks
10. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
11. Adequate hematologic function unless inadequate function is due to underlying disease, such as extensive bone marrow involvement or hypersplenism secondary to the involvement of the spleen by lymphoma per the investigator. Adequate hematologic function is defined as follows:

    o Hemoglobin ≥ 9 g/dL

    o ANC ≥ 1.0 x 10g/L

    o Platelet count ≥ 75 x 10g/L
12. For women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea and age > 45 years) or surgically sterile (absence of ovaries and/or uterus): agreement to remain abstinent or to use single highly effective or combined contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for ≥ 12 months after the last dose of rituximab.

    * Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    * Examples of highly effective contraceptive methods with a failure rate of < 1% per year include tubal ligation, male sterilization, hormonal implants, established, proper use of combined oral or injected hormonal contraceptives, and certain intrauterine devices. Alternatively, two methods (e.g., two barrier methods such as a condom and a cervical cap) may be combined to achieve a failure rate of < 1% per year. Barrier methods must always be supplemented with the use of a spermicide.
13. For women of childbearing potential, a negative serum pregnancy test result within 7 days prior to commencement of dosing. Women who are considered not to be of childbearing potential are not required to have a pregnancy test.
14. For men, agreement to remain abstinent or to use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 6 months after the last dose of study drug and agreement to refrain from donating sperm during this same period.

    * Men with a pregnant partner must agree to remain abstinent or to use a condom for the duration of the pregnancy.
    * Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    * Male patients considering preservation of fertility should bank sperm before treatment with polatuzumab vedotin.

Exclusion Criteria:

1. History of severe allergic or anaphylactic reactions to humanized or murine MAbs (or recombinant antibody-related fusion proteins) or known sensitivity or allergy to murine products
2. Contraindication to bendamustine or rituximab.
3. History of sensitivity to mannitol (mannitol is an excipient in bendamustine).
4. Prior use of any monoclonal antibody (MAb), radioimmunoconjugate, or antibody drug conjugate (ADC) within 5 half-lives or 4 weeks, whichever is longer, before Cycle 1 Day 1.
5. Treatment with chemotherapy, immunotherapy, immunosuppressive therapy, or any investigational agent for the purposes of treating cancer within 2 weeks prior to Cycle 1 Day 1. Radiotherapy for palliative relief of symptoms is allowed.
6. All acute, clinically significant treatment-related toxicity from prior therapy, except for alopecia, must have resolved to Grade ≤ 2 prior to Cycle 1 Day 1.
7. Ongoing corticosteroid use > 30 mg/day prednisone or equivalent, for purposes other than lymphoma symptom control. Patients receiving corticosteroid treatment ≤ 30 mg/day prednisone or equivalent must be documented to be on a stable dose prior to study enrollment and initiation of therapy (Cycle 1 Day 1).
8. Ineligibility for ASCT (determined by investigator per local institutional practice)
9. Prior ASCT
10. History of transformation of indolent disease to DLBCL
11. Active CNS lymphoma. (Previously treated CNS disease is allowed)
12. Current Grade > 1 peripheral neuropathy
13. History of other malignancy that could affect compliance with the protocol or interpretation of results. Exceptions include, but are not limited to:

    • Patients with a history of curatively treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix or ductal carcinoma in situ of the breast at any time prior to the study are eligible.

    • A patient with any other malignancy that has been treated with curative intent and the malignancy has been in remission without treatment for > 3 years prior to enrollment is eligible.

    • Patients with low-grade, early-stage prostate cancer with no requirement for systemic therapy at any time prior to study are eligible.
14. Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results, including significant cardiovascular disease (such as New York Heart Association Class III or IV cardiac disease, myocardial infarction within the last 6 months, unstable arrhythmias, or unstable angina) or significant pulmonary disease (including obstructive pulmonary disease and history of bronchospasm).
15. Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment or any major episode of infection requiring treatment with intravenous (IV) antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior to Cycle 1 Day 1.
16. Patients with suspected or latent tuberculosis. • Latent tuberculosis should be confirmed according to local testing requirements.
17. Positive test results for chronic hepatitis B virus (HBV) infection (defined as positive hepatitis B surface antigen [HBsAg] serology).

    • Patients with occult or prior HBV infection (defined as negative HBsAg and positive hepatitis B core antibody [HBcAb]) may be included if HBV DNA is undetectable, provided that they are willing to undergo DNA testing on day 1 of every cycle and monthly for at least 12 months after the last cycle of study treatment and are willing to get prophylaxis with lamuvidine or entecavir for 6 months post immunosuppressive therapy. Patients who have protective titers of hepatitis B surface antibody (HBsAb) after vaccination or prior but cured hepatitis B are eligible.
18. Patients who are positive for Hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV RNA.
19. Positive test results for uncontrolled HIV infection.

    • For patients with controlled HIV status (Positive HIV antibody, on Antiretroviral therapy with stable HIV viral load) are eligible.
20. Known infection human T-cell leukemia virus 1 (HTLV-1) virus. 21. Vaccination with a live vaccine within 28 days prior to treatment.

22. Recent major surgery (within 6 weeks before the start of Cycle 1 Day 1) other than for diagnosis.

23. Women who are pregnant or lactating or who intend to become pregnant within a year of the last dose of study treatment in the rituximab cohorts or within 18 months of the last dose of study treatment in the obinutuzumab cohort

24. Any of the following abnormal laboratory values, unless abnormal laboratory values are due to underlying lymphoma per the investigator:

* Creatinine > 1.5 x upper limit of normal (ULN) or a measured creatinine clearance < 40 mL/min • AST or ALT > 2.5 x ULN
* Total bilirubin ≥ 1.5 x ULN. Patients with documented Gilbert disease may be enrolled if total bilirubin is ≤ 3 x ULN
* INR or PT > 1.5 x ULN in the absence of therapeutic anticoagulation
* PTT or aPTT > 1.5 x ULN in the absence of a lupus anticoagulant

  25. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Complete response at primary response | 3 weeks after last dose of study medication
  The assessment is based on PET/CT, as determined by the investigator
objective response at primary response | 3 weeks after last dose of study medication
  assessment based on PET/CT as determined by the investigator
duration of response (DOR) of combination therapy | 2 years of follow up
  DOR, defined as the time from the date of the first occurrence of a documented CR or PR to the date of disease progression, relapse, or death from any cause based on PET/CT or CT only as determined by the investigator assessment.Response assessment will be determined according to Modified Lugano Response Criteria for Malignant Lymphoma (Lugano Classification)
number of patients who underwent an ASCT | 2 years of follow up
  Determined during follow up
Cell of Origin analysis | 2 years of follow up
  Cell of origin analysis will be based on immunohistochemistry analysis
Differences in response rates based on timing of relapse | 2 years of follow up
  <12 months of front-line R-chemotherapy versus >12 months after front-line R-chemotherapy and bulky disease prior to ASCT (bulk defined as mass > 7.5 cms)
c-Myc status | 2 years of follow up
  by FISH
2-yr progression free survival (PFS) | 2 years of follow up
  PFS, defined as the time from date of first treatment to the first occurrence of progression or relapse, or death from any cause, based on PET/CT or CT only as determined by the investigator assessment
overall survival (OS) | 2 years of follow up
  defined as the time from the date of randomization or first treatment to the date of death from any cause
stem cell collection failure rate | 2 years of follow up
  Stem cells will be collected post primary response assessment. If patients achieve a PR after 3 cycles of Pola+BR and investigator decides to give additional cycles of Pola+BR (up to a max of 6 cycles) then stem cell collection may occur between cycles to minimize the chances of collection failure.

CONTACTS AND LOCATIONS:
Overall Officials: Brad Haverkos, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No